CLINICAL TRIAL: NCT04686591
Title: A Phase I, Open-label Study of Absolute Bioavailability and Absorption-Distribution-Metabolism-Excretion (ADME) of [14C]AZD9977 in Healthy Male Subjects
Brief Title: Absolute Bioavailability and ADME Study of [14C]AZD9977 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D6402C00002
Record Dates: First submitted 2020-12-17; First posted 2020-12-29 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Disease
Keywords: Chronic Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD9977

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD9977 (Experimental): In Period 1, one 100 mg dose of AZD9977 capsule 50 mg (as 2 x 50 mg capsules) and one 100 µg dose of [14C]AZD9977 Solution for Infusion, 20 µg/mL (NMT 37.0 kBq/5 mL).
  In Period 2, one 100 mg dose of [14C]AZD9977 Oral Suspension, 100 mg (NMT 9.9 MBq).
  Interventions: Drug: AZD9977 capsule 50 mg; Drug: [14C]AZD9977 Solution for Infusion, 20 µg/mL (NMT 37.0 kBq/5 mL); Drug: [14C]AZD9977 Oral Suspension, 100 mg (NMT 9.9 MBq)

INTERVENTIONS:
Drug: AZD9977 capsule 50 mg — 100 mg dose of AZD9977 capsule 50 mg (as 2 x 50 mg capusles)
  Other Names: AZD9977
Drug: [14C]AZD9977 Solution for Infusion, 20 µg/mL (NMT 37.0 kBq/5 mL) — One 100 µg dose of [14C]AZD9977 Solution for Infusion, 20 µg/mL (NMT 37.0 kBq/5 mL)
  Other Names: [14C]AZD9977
Drug: [14C]AZD9977 Oral Suspension, 100 mg (NMT 9.9 MBq) — One 100 mg dose of [14C]AZD9977 Oral Suspension, 100 mg (NMT 9.9 MBq)
  Other Names: [14C]AZD9977

SUMMARY:
Study to Assess the Absorption, Metabolism, and Excretion of [14C]AZD9977 after a Single-Dose Oral Administration

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 30 to 60 years at the time of signing informed consent with suitable veins for cannulation or repeated venepuncture.
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 (body weight at least 50 kg), as measured at screening.
4. Must be willing and able to communicate and participate in the whole study.
5. Must have regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day).
6. Must agree to adhere to the contraception requirements defined in the clinical protocol

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Clinically significant history of recent depression, seizures or other hyperactive central nervous system condition or ongoing treatment for the same.
4. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD9977 or the formulation excipients. Hay fever is allowed unless it is active.
5. Acute diarrhoea or constipation in the 7 days before administration of IMP in the study. If screening occurs >7 days before the first study day, this criterion will be determined on the first study day.
6. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
7. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator.
8. Serum potassium >5.0 mmol/L or fasting blood glucose > upper limit of normal (ULN) at screening.
9. Evidence of renal impairment at screening, as indicated by an estimated eGFR of <80 mL/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation or other evidence of renal impairment.
10. Subjects with known Gilbert's Syndrome or elevated unconjugated hyperbilirubinaemia or subjects with a history of cholecystectomy or gall stones.
11. Abnormal resting vital signs (after 5 min rest) of supine systolic BP >140 mmHg and/or diastolic BP >90 mmHg and/or <50 mmHg and/or HR <45 or >90 bpm at screening or Period 1 Day 1 pre-dose. Vital signs can be repeated once if abnormal, as judged by the investigator.
12. Subjects with clinically significant history of recurrent syncope/blackouts or previous history of orthostatic hypotension or those who are noted to have a fall in systolic BP ≥20 mmHg or diastolic BP ≥10 mmHg or elevation in HR of more than 30 bpm when checked between 2 and 5 min after change of posture at screening or at Period 1 Day 1 pre-dose.
13. Any clinically significant abnormalities on 12-lead ECG, including those which can increase the risk of arrhythmias including QTcF>450 msec, as judged by the investigator.
14. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), and human immunodeficiency virus (HIV) antibody.
15. Known or suspected history of drug abuse in the past 2 years, as judged by the investigator.
16. Has received another new chemical entity (defined as a compound which has not been approved for marketing; including radiolabelled chemical entity) within 90 days of Day 1 in this study. The period of exclusion lasts for 90 days after the final dose or 1 month after the last visit whichever is the longest. Note: subjects consented and screened, but not administered IMP in this study or a previous Phase I study, are not excluded.
17. Involvement of any AstraZeneca, Quotient Sciences or study site employee or their close relatives.
18. Subjects who report to have previously received AZD9977.
19. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
20. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 6 months prior to screening. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
21. Positive screen for drugs of abuse at screening or admission to the clinical unit or confirmed positive alcohol breath test at screening or admission to the clinical unit.
22. Known or suspected history of alcohol abuse or excessive intake of alcohol >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
23. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g., >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
24. Use of any prescribed or non-prescribed medication including antacids, histamine receptor 2 (H2) antagonists, proton pump inhibitors and analgesics (other than up to 4 g paracetamol/acetaminophen per day), herbal remedies (including but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto and ginseng), megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to the first administration of IMP or longer if the medication has a long half-life. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
25. Evidence of current SARS-CoV-2 infection.
26. Subjects with pregnant or lactating partners.
27. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
28. Subjects who have been administered IMP in an 14C ADME study in the last 12 months.
29. Subjects who cannot communicate reliably with the investigator.
30. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
31. Judgment by the investigator that the volunteer should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
32. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of AZD9977 | Collection of plasma samples from pre-dose until 72 hours post-dose.
  Absolute bioavailability based on AUC0-inf of oral formulation compared to IV adjusted for dose
The cumulative amount of AZD9977 excreted (CumAe) | Collection of urine and faecal samples from pre-dose until 168 hours post-dose.
  Assessment of the total radioactivity by measuring the cumulative amount of AZD9977 excreted (CumAe)
The cumulative amount of AZD9977 excreted and expressed as a percentage of the administered dose (CumFe) | Collection of urine and faecal samples from pre-dose until 168 hours post-dose.
  Assessment of the rates and routes of elimination by measuring the cumulative amount excreted and expressed as a percentage of the administered dose (CumFe)
Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of plasma samples from pre-dose until 72 hours post-dose in period 1 and from pre-dose to 168 hours post-dose in period 2.
  Assessment of metabolites in plasma by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of urine samples from pre-dose until 72 hours post-dose in period 1 and from pre-dose to 168 hours post-dose in period 2.
  Assessment of metabolites in urine by liquid chromatography-radiochemical-detection and subsequent mass spectrometry
Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry | Collection of faecal samples from pre-dose until 168 hours post-dose.
  Assessment of metabolites in faeces by liquid chromatography-radiochemical-detection and subsequent mass spectrometry

SECONDARY OUTCOMES:
Number of adverse events (AEs) experienced by subjects | Approximately 8 weeks
  Safety and tolerability assessed through the incidence of AEs
Time prior to the first measurable concentration (AZD9977) (tlag) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring the time to first measurable concentration (tlag)
Time of maximum observed concentration (tmax) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring time of maximum observed concentration (tmax)
Maximum observed concentration (cmax) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring maximum observed concentration (cmax)
Area under the curve from time 0 to the time of last measurable concentration (AUC0-t) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring area under the curve from time 0 to the time of last measurable concentration (AUC0-t)
Area under the curve from time 0 extrapolated to infinity (AUC0-inf) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 by measuring area under the curve from time 0 extrapolated to infinity (AUC0-inf)
Area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC%extrap) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring area under the curve from time of the last measurable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC%extrap)
Terminal half-life (t1/2) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring terminal half-life (t1/2)
First order rate constant associated with the terminal (log-linear) portion of the curve (λz) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 and total radioactivity by measuring first order rate constant associated with the terminal (log-linear) portion of the curve (λz)
Total body clearance calculated after a single oral administration (AZD9977) (CL/F) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 by measuring total body clearance calculated after a single oral administration (AZD9977) (CL/F)
Renal clearance calculated using plasma AUC (AZD9977 and [14C]AZD9977) (CLr) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 by measuring Renal clearance calculated using plasma AUC (AZD9977 and [14C]AZD9977) (CLr)
Apparent volume of distribution based on the terminal phase calculated using AUC0 inf after a single oral administration (AZD9977) (Vz/F) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 by measuring apparent volume of distribution based on the terminal phase calculated using AUC0 inf after a single oral administration (AZD9977) (Vz/F)
Mean residence time from time 0 to time of the last measurable concentration (AZD9977 and [14C]AZD9977) (MRT0-t) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 by measuring mean residence time from time 0 to time of the last measurable concentration (AZD9977 and [14C]AZD9977) (MRT0-t)
Mean residence time extrapolated to infinity (AZD9977 and [14C]AZD9977) (MRT0-inf) | Collection of plasma samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of pharmacokinetics of AZD9977 and [14C]AZD9977 by measuring mean residence time extrapolated to infinity (AZD9977 and [14C]AZD9977) (MRT0-inf)
Total body clearance calculated after a single intravenous administration ([14C]AZD9977) (CL) | Collection of plasma samples from pre-dose to 72 hours post-dose
  Assessment of pharmacokinetics of [14C]AZD9977 by measuring total body clearance calculated after a single intravenous administration ([14C]AZD9977) (CL)
Volume of distribution at steady state after a single intravenous administration ([14C]AZD9977) (Vss) | Collection of plasma samples from pre-dose to 72 hours post-dose
  Assessment of pharmacokinetics of [14C]AZD9977 by measuring volume of distribution at steady state after a single intravenous administration ([14C]AZD9977) (Vss)
Volume of distribution based on the terminal phase calculated using AUC0 inf after a single intravenous administration ([14C]AZD9977) (Vz | Collection of plasma samples from pre-dose to 72 hours post-dose
  Assessment of pharmacokinetics of [14C]AZD9977 by measuring volume of distribution based on the terminal phase calculated using AUC0 inf after a single intravenous administration ([14C]AZD9977) (Vz)
Evaluation of whole blood:plasma concentration ratios for total radioactivity | Collection of blood samples from pre-dose to 72 hours post-dose in period 1 and pre-dose to 168 hours post-dose in period 2.
  Assessment of total radioactivity in whole blood and plasma

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  URL:
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home